CLINICAL TRIAL: NCT00292591
Title: Evaluation of Vitamin D Requirements During Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Carol Wagner, Professor of Pediatrics, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R01HD043921 (NIH); 5R01HD043921 (NIH)
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-08

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; cholecalciferol; pregnancy; bone mineral density
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- cholecalciferol-400 IU (Active Comparator): Control group receiving 400 IU/day plus 0 IU vitamin D3 as placebo/day
  Interventions: Drug: cholecalciferol (vitamin D3); Drug: cholecalciferol
- cholecalciferol 2000 IU (Experimental): Experimental group receiving 2000 IU total vitamin D3/day.
  Interventions: Drug: cholecalciferol (vitamin D3); Drug: cholecalciferol
- cholecalciferol 4000 IU (Experimental): Experimental group receiving 4000 IU/day cholecalciferol
  Interventions: Drug: cholecalciferol (vitamin D3); Drug: cholecalciferol

INTERVENTIONS:
Drug: cholecalciferol (vitamin D3) — randomized control trial of three vitamin D doses: 400, 2000 and 4000 IU/day
Drug: cholecalciferol — comparing vitamin D requirements of pregnant women and their fetuses from 12 weeks' gestation through pregnancy
  Other Names: vitamin D3

SUMMARY:
The purpose of this study is to determine the effectiveness of vitamin D supplementation during pregnancy starting at the beginning of the second trimester. Mothers will be randomized to one of three vitamin D dosing groups: 400, 2,000 or 4,000 international units per day. It is hypothesized that the highest dosing regimen will result in a better vitamin D status of women regardless of their ethnicity or race.

DETAILED DESCRIPTION:
The prevalence of hypovitaminosis D in reproductive aged African-American women occurs at a rate of > 40%. Two factors have contributed to this public health problem: an inadequate DRI for vitamin D and avoidance of sun exposure/use of sunscreen. This startling rate of hypovitaminosis D requires that the DRI for vitamin D in pregnancy be evaluated in a detailed manner. The Cochrane Library (2002) released a report stating that there is insufficient data to evaluate the effects of vitamin D supplementation during pregnancy. Recently, the safety of prolonged supplementation with up to 25x's DRI (10,000 IU/day) was demonstrated in nonpregnant adults. It is essential to determine what dose of vitamin D is required to eliminate hypovitaminosis D during pregnancy and provide the fetus/neonate with adequate vitamin D stores during development and growth, particularly in darkly pigmented individuals. The aim of this research proposal, then, is to determine the efficacy, effectiveness, and safety of maternal vitamin D supplementation (as a function of ethnicity and UV exposure) in the prevention of hypovitaminosis D in the pregnant mother and her fetus/neonate. We hypothesize that darkly pigmented mothers will require substantially higher oral supplementation with vitamin D to eliminate hypovitaminosis D as compared to their Caucasian counterparts. We propose a comprehensive clinical trial to test our hypothesis. Mothers at 12 weeks' gestation will be randomized to one of three vitamin D treatment groups:

1. Control, 400-,
2. 2,000-, or
3. 4,000 IU/day to be continued throughout pregnancy.

Calcium and vitamin D homeostasis and skeletal remodeling in the mother will be monitored closely throughout the pregnancy. Bone density of the mother will be measured at 12 weeks' gestation and one-month postpartum. Follow-up growth and skeletal integrity assessments of the infant will be performed at birth, 1, 6 and 12 months stratified by infant feeding regime. Through these proposed studies, the prevalence of hypovitaminosis D among mothers, their developing fetuses and neonates, and the utility of maternal therapeutic intervention with vitamin D for both mother and fetus/infant will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are within the ages of 16-45 years
2. In good general health
3. Less than 12 weeks pregnant (based on last menstrual period)

Exclusion Criteria:

1. Mothers with preexisting type I or type II diabetes
2. Mothers with preexisting hypertension
3. Mothers with preexisting parathyroid disease or uncontrolled thyroid disease
4. Mothers with multiple fetuses (e.g., twins, triplets, etc.)

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 501 (Actual)
Dates: Start 2004-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce W. Hollis, Ph.D., Principal Investigator — Medical University of South Carolina; Carol L. Wagner, M.D., Principal Investigator — Medical University of South Carolina; Donna Johnson, M.D., Study Director — Medical University of South Carolina; Thomas C. Hulsey, Sc.D., Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Hollis BW. Circulating 25-hydroxyvitamin D levels indicative of vitamin D sufficiency: implications for establishing a new effective dietary intake recommendation for vitamin D. J Nutr. 2005 Feb;135(2):317-22. doi: 10.1093/jn/135.2.317. PMID 15671234
- [Background] Hollis BW, Wagner CL. Normal serum vitamin D levels. N Engl J Med. 2005 Feb 3;352(5):515-6; author reply 515-6. doi: 10.1056/NEJM200502033520521. No abstract available. PMID 15689596
- [Result] Hollis BW, Johnson D, Hulsey TC, Ebeling M, Wagner CL. Vitamin D supplementation during pregnancy: double-blind, randomized clinical trial of safety and effectiveness. J Bone Miner Res. 2011 Oct;26(10):2341-57. doi: 10.1002/jbmr.463. Erratum In: J Bone Miner Res. 2011 Dec; 26(12):3001. PMID 21706518
- [Result] Hollis BW, Wagner CL. Vitamin D requirements and supplementation during pregnancy. Curr Opin Endocrinol Diabetes Obes. 2011 Dec;18(6):371-5. doi: 10.1097/MED.0b013e32834b0040. PMID 21857221
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] Wei W, Shary JR, Garrett-Mayer E, Anderson B, Forestieri NE, Hollis BW, Wagner CL. Bone mineral density during pregnancy in women participating in a randomized controlled trial of vitamin D supplementation. Am J Clin Nutr. 2017 Dec;106(6):1422-1430. doi: 10.3945/ajcn.116.140459. Epub 2017 Oct 18. PMID 29046301

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cholecalciferol-400 IU | Cholecalciferol 2000 IU | Cholecalciferol 4000 IU
Started | 166 | 167 | 168
Completed | 102 | 111 | 110
Not Completed | 64 | 56 | 58

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cholecalciferol-400 IU | Cholecalciferol 2000 IU | Cholecalciferol 4000 IU | Total
Number analyzed (Participants) | 166 | 167 | 168 | 501
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (5.6) | 26.7 (5.5) | 26.4 (5.4) | 26.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 167 | 168 | 501
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 25-Hydroxyvitamin D Concentration
Description: Circulating total 25(OH)D concentration measured in serum at visit 7, one month prior to delivery
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cholecalciferol-400 IU | Cholecalciferol 2000 IU | Cholecalciferol 4000 IU
Number analyzed (Participants) | 102 | 111 | 110
ng/mL | 32.5 (14.4) | 41.0 (14.6) | 45.7 (14.3)

ADVERSE EVENTS:
Arm/Group | Cholecalciferol-400 IU | Cholecalciferol 2000 IU | Cholecalciferol 4000 IU
Serious Adverse Events (participants affected / at risk) | 9/166 | 4/167 | 13/168
Other Adverse Events (participants affected / at risk) | 22/166 | 35/167 | 27/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholecalciferol-400 IU (N=166) | Cholecalciferol 2000 IU (N=167) | Cholecalciferol 4000 IU (N=168)
Pregnancy loss (miscarriage/fetal death) (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 4 (4) | 13 (13)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholecalciferol-400 IU (N=166) | Cholecalciferol 2000 IU (N=167) | Cholecalciferol 4000 IU (N=168)
Complications of Pregnancy (Pregnancy, puerperium and perinatal conditions) | 22 (22) | 35 (35) | 27 (27) — Examples include preterm birth or labor complications due to infection, pre-eclampsia, gestational diabetes, etc. (not reported separately due to small numbers)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No